CLINICAL TRIAL: NCT04228679
Title: The Affect of Erbium Laser Treatments on Vaginal Looseness and Sexual Dysfunction in Pre-menopausal Female Individuals.
Brief Title: Erbium Laser for Treatment of Vaginal Looseness and Sexual Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0309-19-RMB
Record Dates: First submitted 2020-01-12; First posted 2020-01-14 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erbium laser treatment (Experimental): Women with vaginal looseness and sexual dysfunction treated with real laser.
  Interventions: Device: Erbium laser
- Sham laser treatment (Sham Comparator): Women with vaginal looseness and sexual dysfunction treated with sham laser.
  Interventions: Device: Sham Laser

INTERVENTIONS:
Device: Erbium laser — Erbium laser device
  Arms: Erbium laser treatment
Device: Sham Laser — Sham laser device
  Arms: Sham laser treatment

SUMMARY:
Patients with a primary complaint of vaginal looseness and sexual dysfunction, visiting a sexual dysfunction clinic at a tertiary medical center will undergo randomization to either a series of 3 laser treatments or 3 sham treatments, and the effect of these treatments will be measured by several validated questionaires and by means of gynecological examination.

DETAILED DESCRIPTION:
Patients suffering from vaginal looseness and sexual dysfunction, as a primary sexual dysfunction complaint will be recruited, sign an informed consent and will receive a thorough explanation regarding the side effects and possible beneficial affects the laser treatments may bestow.

Patients will undergo randomization to either a series of 3 laser treatments or 3 sham treatments, and the effect of these treatments will be measured by several validated questionaires and by means of gynecological examination.

Follow up after treatment cessation will be for 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women.
* Women with vaginal looseness and sexual dysfunction as a primary complaint.

Exclusion Criteria:

* Vaginal bleeding of unknown source.
* Repeated vaginal infections.
* Known or suspected cervical pre-malignant neoplasia.
* Previous treatment with vaginal laser or other forms of energy-based treatment modalities.
* Pregnancy.
* Current pelvic inflammatory disease or urinary tract infection.
* Vaginal surgery during the year preceding study participation.
* Treatment with systemic or vaginal hormone replacement therapy.
* Current pelvic floor physiotherapy.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 106 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Female sexual function index. | From recruitment up to 15 months.
  Female sexual function index scores pre- and post-treatment. Minimal score is 2, maximal score is 36. Thee higher the score, the improved the sexual function is.

SECONDARY OUTCOMES:
Vaginal health index | From recruitment up to 15 months.
  Vaginal health index score. The total VHI scores range between 5 and 25. A higher score indicates increased vaginal health.
Pelvic floor disability index. | From recruitment up to 15 months.
  Changes in the pelvic floor disability index scores pre- and post-treatment. Minimal score is 0, maximal score is 300. The higher the score, the improved the worse pelvic floor dysfunction is.
Vaginal laxity questionnaire. | From recruitment up to 15 months.
  Changes in the vaginal laxity questionnaire scores pre- and post-treatment. Minimal score is 1, maximal score is 7. The lower the score, the worse vaginal laxity is.
Monthly sexual intercourse rate | From recruitment up to 15 months.
  Average monthly sexual intercourse rates.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No